CLINICAL TRIAL: NCT02982954
Title: Phase 3b/4 Safety Trial of Nivolumab Combined With Ipilimumab in Subjects With Previously Untreated, Advanced or Metastatic RCC (CheckMate 920: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 920)
Brief Title: A Study to Evaluate the Safety of Nivolumab and Ipilimumab in Subjects With Previously Untreated Advanced or Metastatic Renal Cell Cancer
Acronym: CHECKMATE 920
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-920
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ccRCC KPS ≥ 70% (Experimental): Clear-Cell Renal Cell Carcinoma (ccRCC) with Karnofsky Performance Status (KPS) ≥ 70%
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Non-ccRCC, KPS ≥ 70% (Experimental): Non Clear-Cell Renal Cell Carcinoma (nccRCC) with KPS ≥ 70%
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- RCC with non-active Brain Mets, KPS ≥70% (Experimental): Renal Cell Carcinoma (RCC) with non-active Brain Metastases, with KPS ≥70%
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- any RCC with KPS 50%-60% (Experimental): Renal Cell Carcinoma (RCC), regardless of any histology or existing non-active brain metastasis, with KPS 50%-60%
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified day
  Other Names: BMS-936558; Opdivo
Drug: Ipilimumab — Specified Dose on Specified Day
  Other Names: Yervoy; BMS-734016

SUMMARY:
To investigate the safety of Nivolumab in combination with Ipilimumab in subjects with previously untreated advanced or metastatic Renal Cell Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Type of Participant and Target Disease Characteristics

1. Advanced or metastatic RCC
2. Histologically confirmed, previously untreated (treatment-naive) RCC
3. No prior systemic therapy for RCC except for one prior adjuvant or neoadjuvant therapy for completely resectable RCC
4. Measurable disease as per RECIST 1.1. Subject must have extracranial metastasis as measurable disease
5. Karnofsky Performance Status (KPS) of at least 70% for Cohort 1, 2, and 3; KPS of 50-60% for Cohort 4
6. Tumor tissue need be received by the central vendor (block or unstained slides). Note: Fine Needle Aspiration (FNA)and bone metastases samples are not acceptable for submission.

Exclusion Criteria:

1. Medical Conditions

   1. Subjects with any active autoimmune disease or a history of known autoimmune disease
   2. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured
   3. Known HIV or AIDS-related illness
   4. Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection.
2. Prior/Concomitant Therapy

   1. Prior systemic treatment in the metastatic setting with Vascular epithelial growth factor(VEGF) or VEGF receptor targeted therapy
   2. Prior treatment with an anti-Programmed Death (PD) -1, anti-PD-L1, anti-PD-L2, anti-cluster of differentiation 137 (CD137), or anti-cytotoxic T-lymphocyte-associated antigen 4(CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways. This includes the utilization of these agents in the neo-adjuvant or adjuvant setting.
   3. Anti-cancer therapy less than 28 days prior to the first dose of study drug or palliative, focal radiation therapy less than 14 days prior to the first dose of study drug.

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (61):
- United States (61):
  - Northwest Alabama Cancer Center, Pc, Muscle Shoals, Alabama
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Ironwood Cancer And Research Centers, Pc, Chandler, Arizona
  - Local Institution - 0028, Fayetteville, Arkansas
  - eCare, Encinitas, California
  - Pacific Shores Medical Group, Long Beach, California
  - Los Angeles Cancer Network, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - Torrance Health Association, Redondo Beach, California
  - Kaiser Permanente Medical Group - Southern California, Riverside, California
  - Sharp Memorial Hospital, San Diego, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Med Oncology, Santa Maria, California
  - Florida Cancer Specialists S., Fort Myers, Florida
  - University Of Miami/Sylvester Cancer Center, Miami, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - Local Institution - 0012, Fort Wayne, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Southdale Cancer Clinic, Burnsville, Minnesota
  - Local Institution - 0009, Coon Rapids, Minnesota
  - Park Nicollet Clinic Cancer Center, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - HCA Midwest Division, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Local Institution - 0023, Hackensack, New Jersey
  - University Of New Mexico, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - St. Francis Cancer Treatment Center, Grand Island, New York
  - Broome Oncology, Johnson City, New York
  - Local Institution - 0052, New York, New York
  - Weill Cornell Medical College, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oklahoma Cancer Specialists and Research Institute, LLC-Clinical Research, Tulsa, Oklahoma
  - Local Institution - 0071, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - Hollings Cancer Center, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC - SCRI - PPDS, Chattanooga, Tennessee
  - Local Institution - 0002, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-Fort Worth 12th Ave, Fort Worth, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Local Institution - 0042, Fairfax, Virginia
  - Bon Secours St Francis Hospital, Midlothian, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

REFERENCES:
- [Derived] George DJ, Spigel DR, Gordan LN, Kochuparambil ST, Molina AM, Yorio J, Rezazadeh Kalebasty A, McKean H, Tchekmedyian N, Tykodi SS, Zhang J, Askelson M, Johansen JL, Hutson TE. Safety and efficacy of first-line nivolumab plus ipilimumab alternating with nivolumab monotherapy in patients with advanced renal cell carcinoma: the non-randomised, open-label, phase IIIb/IV CheckMate 920 trial. BMJ Open. 2022 Sep 14;12(9):e058396. doi: 10.1136/bmjopen-2021-058396. PMID 36104138
- [Derived] Tykodi SS, Gordan LN, Alter RS, Arrowsmith E, Harrison MR, Percent I, Singal R, Van Veldhuizen P, George DJ, Hutson T, Zhang J, Zoco J, Johansen JL, Rezazadeh Kalebasty A. Safety and efficacy of nivolumab plus ipilimumab in patients with advanced non-clear cell renal cell carcinoma: results from the phase 3b/4 CheckMate 920 trial. J Immunother Cancer. 2022 Feb;10(2):e003844. doi: 10.1136/jitc-2021-003844. PMID 35210307
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Nivolumab 6mg/kg IV plus, Ipilimumab 1mg/kg IV every 8 weeks alternating with Nivolumab 480 mg IV every 8 weeks, staggered every 4 weeks
- Cohort 2; Cohort 3: Nivolumab 3mg/kg IV combined with Ipilimumab 1mg/kg IV every 3 weeks for 4 doses
- Cohort 4: Nivolumab 3 mg/kg IV combined with Ipilimumab 1 mg/kg IV every 3 weeks for 4 doses
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 106 | 52 | 28 | 25
Completed | 0 | 0 | 0 | 0
Not Completed | 106 | 52 | 28 | 25
Not completed — Death | 55 | 29 | 15 | 20
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Participant withdrew consent | 7 | 5 | 1 | 1
Not completed — Other reasons | 42 | 17 | 12 | 3
Not completed — Premature site closure | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 106 | 52 | 28 | 25 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (9.43) | 60.1 (14.09) | 61.3 (11.06) | 65.2 (12.54) | 62.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 4 | 6 | 46
  Male | 86 | 36 | 24 | 19 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 1 | 1 | 10
  Not Hispanic or Latino | 101 | 48 | 27 | 24 | 200
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 1 | 1 | 9
  White | 104 | 40 | 26 | 24 | 194
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Grade (Grade 3-4) Immune Mediated Adverse Events (IMAEs)
Description: Number of participants with IMAEs in the following categories: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity
Time Frame: Approximately 39 Months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Participants
  Pneumonitis | 1 | 0 | 0 | 0
  Diarrhoea/Colitis | 8 | 4 | 2 | 0
  Hepatitis | 3 | 1 | 1 | 1
  Nephritis and Renal Dysfunction | 0 | 2 | 0 | 0
  Rash | 7 | 3 | 1 | 0
  Hypersensitivity | 0 | 0 | 0 | 0
  Adrenal Insufficiency | 3 | 1 | 0 | 1
  Hypothyroidism and Thyroiditis | 0 | 0 | 0 | 1
  Diabetes Mellitus | 3 | 0 | 1 | 0
  Hyperthyroidism | 0 | 0 | 0 | 0
  Hypophysitis | 0 | 1 | 1 | 0

2. Primary Outcome: Number of Participants With High Grade (Grade 5) Immune Mediated Adverse Events (IMAEs)
Description: as for outcome 1
Time Frame: Approximately 39 Months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Participants
  Pneumonitis | 0 | 0 | 0 | 0
  Diarrhoea/Colitis | 0 | 0 | 0 | 0
  Hepatitis | 0 | 0 | 0 | 0
  Nephritis and Renal Dysfunction | 0 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 0
  Hypersensitivity | 0 | 0 | 0 | 0
  Adrenal Insufficiency | 0 | 0 | 0 | 0
  Hypothyroidism and Thyroiditis | 0 | 0 | 0 | 0
  Diabetes Mellitus | 0 | 0 | 0 | 0
  Hyperthyroidism | 0 | 0 | 0 | 0
  Hypophysitis | 0 | 0 | 0 | 0

3. Secondary Outcome: Time to Onset of Grade 3-5 Immune Mediated Adverse Events (IMAEs)
Description: Time to onset is defined as the duration of time in weeks from the first dosing to the immune modulating adverse event onset date. Participants experiencing all high grade (CTCAE v4 Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs) in the following categories will be included: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity. IMAEs are specific events (or groups of preferred terms describing specific events) considered as potential immune-mediated events by investigator, that meet the following definition: (1) those occurring within 100 days of the last dose (2) regardless of causality (3) with no clear alternate etiology based on investigator assessment, or with an immune-mediated component and (4) treated with immune-modulating medication. Grade 3= Severe reaction, Grade 4 = Life-threatening, Grade 5 = Death
Time Frame: From first dose to the earliest IMAE (grade 3-5) event onset date (up to approximately 116 weeks)
Population: All Treated Participants Who Experienced at Least 1 IMAE Where Immune-modulating Medication was Initiated
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Weeks
  Pneumonitis: number analyzed (Participants) | 1 | 0 | 0 | 0
  Pneumonitis | 12.7 [12.7 to 12.7] |  |  |
  Diarrhoea/Colitis: number analyzed (Participants) | 8 | 4 | 2 | 0
  Diarrhoea/Colitis | 21.79 [1.7 to 115.7] | 10.43 [4.4 to 20.1] | 11.0 [10.1 to 11.9] |
  Hepatitis: number analyzed (Participants) | 3 | 1 | 1 | 1
  Hepatitis | 8.43 [2.0 to 82.1] | 9.4 [9.4 to 9.4] | 11.6 [11.6 to 11.6] | 10.1 [10.1 to 10.1]
  Nephritis and Renal Dysfunction: number analyzed (Participants) | 0 | 2 | 0 | 0
  Nephritis and Renal Dysfunction |  | 9.43 [1.4 to 17.4] |  |
  Rash: number analyzed (Participants) | 7 | 3 | 1 | 0
  Rash | 4.00 [1.1 to 80.4] | 6.14 [2.3 to 13.7] | 8.3 [8.3 to 8.3] |
  Hypersensitivity: number analyzed (Participants) | 0 | 0 | 0 | 0
  Immune Mediated Arthritis: number analyzed (Participants) | 0 | 1 | 0 | 0
  Immune Mediated Arthritis |  | 38.9 [38.9 to 38.9] |  |
  Myositis/Rhabdomyolysis Event: number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal Insufficiency: number analyzed (Participants) | 2 | 1 | 0 | 1
  Adrenal Insufficiency | 36.21 [21.0 to 51.4] | 12.7 [12.7 to 12.7] |  | 14.9 [14.9 to 14.9]
  Hypothyroidism and Thyroiditis: number analyzed (Participants) | 0 | 0 | 0 | 0
  Diabetes Mellitus: number analyzed (Participants) | 0 | 0 | 1 | 0
  Diabetes Mellitus |  |  | 2.0 [2.0 to 2.0] |
  Hyperthyroidism: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hypophysitis |  | 18.7 [18.7 to 18.7] |  |

4. Secondary Outcome: Time to Resolution of Grade 3-5 Immune Mediated Adverse Events (IMAEs)
Description: Time to resolution is defined as the longest time from IMAE onset date to complete resolution or improvement to the grade at baseline experienced by the participant (the IMAE end date). Participants experiencing all high grade (CTCAE v4 Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs) in the following categories will be included: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity. IMAEs are specific events (or groups of preferred terms describing specific events) considered as potential immune-mediated events by investigator, that meet the following definition: (1) those occurring within 100 days of the last dose (2) regardless of causality (3) with no clear alternate etiology based on investigator assessment, or with an immune-mediated component and (4) treated with immune-modulating medication. Grade 3= Severe reaction, Grade 4 = Life-threatening, Grade 5 = Death
Time Frame: From the IMAE onset date to the IMAE end date, up to approximately 194 weeks
Population: All Treated Participants Who Experienced at Least 1 IMAE Where Immune-modulating Medication was Initiated
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Weeks
  Pneumonitis: number analyzed (Participants) | 1 | 0 | 0 | 0
  Pneumonitis | 0.9 [0.9 to 0.9] |  |  |
  Diarrhoea/Colitis: number analyzed (Participants) | 9 | 4 | 3 | 0
  Diarrhoea/Colitis | 2.71 [0.7 to 193.9] | 5.93 [0.9 to 16.9] | 1.14 [1.1 to 4.9] |
  Hepatitis: number analyzed (Participants) | 3 | 2 | 1 | 1
  Hepatitis | NA [7.9 to 144.9] — Median not calculated due to insufficient number of events. | NA [14.9 to 18.3] — Median not calculated due to insufficient number of events. | 3.00 [3.0 to 3.0] | 2.1 [2.1 to 2.1]
  Nephritis and Renal Dysfunction: number analyzed (Participants) | 0 | 2 | 0 | 0
  Nephritis and Renal Dysfunction |  | 7.79 [1.1 to 14.4] |  |
  Rash: number analyzed (Participants) | 7 | 3 | 1 | 0
  Rash | 26.86 [5.3 to 181.6] | 8.00 [3.1 to 69.9] | 5.3 [5.3 to 5.3] |
  Hypersensitivity: number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal Insufficiency: number analyzed (Participants) | 2 | 0 | 0 | 1
  Adrenal Insufficiency | NA [0.4 to 170.0] — Median not calculated due to insufficient number of events. |  |  | 6.0 [6.0 to 6.0]
  Diabetes Mellitus: number analyzed (Participants) | 0 | 0 | 1 | 0
  Diabetes Mellitus |  |  | 1.1 [1.1 to 1.1] |
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hypophysitis |  | 7.6 [7.6 to 7.6] |  |
  Immune Mediated Arthritis: number analyzed (Participants) | 0 | 1 | 0 | 0
  Immune Mediated Arthritis |  | 37.0 [37.0 to 37.0] |  |

5. Secondary Outcome: Number of Participants Who Received Immune Modulating Medication for High Grade (Grades 3-5) Immune Mediated Adverse Events (IMAEs)
Description: The number of participants who received immune modulating medication for participants experiencing all high grade (CTCAE v4 Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs) in the following categories will be included: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity. IMAEs are specific events (or groups of preferred terms describing specific events) considered as potential immune-mediated events by investigator, that meet the following definition: (1) those occurring within 100 days of the last dose (2) regardless of causality (3) with no clear alternate etiology based on investigator assessment, or with an immune-mediated component and (4) treated with immune-modulating medication. Grade 3= Severe reaction, Grade 4 = Life-threatening, Grade 5 = Death
Time Frame: From first dose up to 100 days post last dose (up to approximately 29 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Participants
  Pneumonitis: number analyzed (Participants) | 1 | 0 | 0 | 0
  Pneumonitis | 1 | 0 | 0 | 0
  Diarrhoea/Colitis: number analyzed (Participants) | 8 | 4 | 2 | 0
  Diarrhoea/Colitis | 8 | 4 | 2 | 0
  Hepatitis: number analyzed (Participants) | 3 | 1 | 1 | 1
  Hepatitis | 3 | 1 | 1 | 1
  Nephritis and Renal Dysfunction: number analyzed (Participants) | 0 | 2 | 0 | 0
  Nephritis and Renal Dysfunction | 0 | 2 | 0 | 0
  Rash: number analyzed (Participants) | 7 | 3 | 1 | 0
  Rash | 7 | 3 | 1 | 0
  Hypersensitivity: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hypersensitivity | 0 | 0 | 0 | 0
  Adrenal Insufficiency: number analyzed (Participants) | 3 | 1 | 0 | 1
  Adrenal Insufficiency | 3 | 1 | 0 | 1
  Hypothyroidism/Thyroiditis: number analyzed (Participants) | 0 | 0 | 0 | 1
  Hypothyroidism/Thyroiditis | 0 | 0 | 0 | 1
  Diabetes Mellitus: number analyzed (Participants) | 3 | 0 | 1 | 0
  Diabetes Mellitus | 3 | 0 | 1 | 0
  Hyperthyroidism: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hyperthyroidism | 0 | 0 | 0 | 0
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 1 | 0
  Hypophysitis | 0 | 1 | 1 | 0

6. Secondary Outcome: Number of Participants Who Received Hormone Replacement Therapy for High Grade (Grades 3-5) Immune Mediated Adverse Events (IMAEs)
Description: The number of participants who received Hormone Replacement Therapy for experiencing all high grade (CTCAE v4 Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs) in the following categories will be included: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity. IMAEs are specific events (or groups of preferred terms describing specific events) considered as potential immune-mediated events by investigator, that meet the following definition: (1) those occurring within 100 days of the last dose (2) regardless of causality (3) with no clear alternate etiology based on investigator assessment, or with an immune-mediated component and (4) treated with immune-modulating medication. Grade 3= Severe reaction, Grade 4 = Life-threatening, Grade 5 = Death
Time Frame: From first dose up to 100 days post last dose (up to approximately 29 months)
Population: Treated participants who experienced at least one Grade 3 to 5 Immune-Mediate Event from the category
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Participants
  Pneumonitis: number analyzed (Participants) | 1 | 0 | 0 | 0
  Pneumonitis | 1 | 0 | 0 | 0
  Diarrhoea/Colitis: number analyzed (Participants) | 8 | 4 | 2 | 0
  Diarrhoea/Colitis | 8 | 3 | 2 | 0
  Hepatitis: number analyzed (Participants) | 3 | 1 | 1 | 1
  Hepatitis | 3 | 1 | 1 | 1
  Nephritis and Renal Dysfunction: number analyzed (Participants) | 0 | 2 | 0 | 0
  Nephritis and Renal Dysfunction | 0 | 2 | 0 | 0
  Rash: number analyzed (Participants) | 7 | 3 | 1 | 0
  Rash | 7 | 3 | 1 | 0
  Hypersensitivity: number analyzed (Participants) | 0 | 0 | 0 | 0
  Adrenal Insufficiency: number analyzed (Participants) | 3 | 1 | 0 | 1
  Adrenal Insufficiency | 2 | 1 | 0 | 1
  Hypothyroidism and Thyroiditis: number analyzed (Participants) | 0 | 0 | 0 | 0
  Diabetes Mellitus: number analyzed (Participants) | 3 | 0 | 1 | 0
  Diabetes Mellitus | 0 | 0 | 1 | 0
  Hyperthyroidism: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 1 | 0
  Hypophysitis | 0 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants Who Received ≥ 40mg of Prednisone for High Grade (Grades 3-5) Immune Mediated Adverse Events (IMAEs)
Description: The number of participants who received ≥ 40mg of prednisone for high grade (grades 3-5) IMAEs. Participants experiencing all high grade (CTCAE v4 Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs) in the following categories will be included: Skin, Endocrine, Gastrointestinal, Hepatic, Renal, Pulmonary and Hypersensitivity. IMAEs are specific events (or groups of preferred terms describing specific events) considered as potential immune-mediated events by investigator, that meet the following definition: (1) those occurring within 100 days of the last dose (2) regardless of causality (3) with no clear alternate etiology based on investigator assessment, or with an immune-mediated component and (4) treated with immune-modulating medication. Grade 3= Severe reaction, Grade 4 = Life-threatening, Grade 5 = Death
Time Frame: From first dose up to 100 days post last dose (up to approximately 29 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Participants | 19 | 9 | 5 | 2

8. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose to the date of the first documented progressive disease (PD) as determined by the investigator (per RECIST 1.1 criteria or clinical) or death due to any cause whichever occur first. Progressive disease is defined as progression of existing non-target lesions or at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From first dose to the date of the first documented progressive disease, up to approximately 12 months
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 106 | 52 | 28 | 25
Months | 4.8 [3.0 to 8.4] | 3.7 [2.7 to 4.6] | 8.5 [2.9 to 12.0] | 3.6 [2.5 to 8.7]

9. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable participants. Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment. The participant's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all lesions and normalization of tumor marker level. All lymph nodes (whether target or non-target) must be non-pathological in size (< 10mm short axis).
Time Frame: From first dose up to the date of objectively documented progression or the date of subsequent therapy, whichever occurs first (up to approximately 26 months)
Population: All response evaluable participants: all treated participants who have baseline and at least one on-study evaluable tumor measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 96 | 46 | 26 | 18
Percentage of Participants | 35.4 [25.9 to 45.8] | 21.7 [10.9 to 36.4] | 30.8 [14.3 to 51.8] | 33.3 [13.3 to 59.0]

10. Secondary Outcome: Time to Response Rate (TRR)
Description: TTR is defined as the median percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable participants. Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment. The participant's best overall response assignment will depend on the findings of both target and non-target disease and will also take into consideration the appearance of new lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all lesions and normalization of tumor marker level. All lymph nodes (whether target or non-target) must be non-pathological in size (< 10mm short axis).
Time Frame: From the date of first dose to first documented CR or PR, up to approximately 15 months
Population: as for outcome 9
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 96 | 46 | 26 | 18
Months | 2.8 [2.5 to 14.6] | 2.8 [2.1 to 4.5] | 2.8 [2.4 to 3.0] | 4.5 [2.5 to 12.1]

11. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time between the date of first confirmed response to the date of the first documented tumor progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, or death due to any cause, whichever occurs first. DOR will be computed for participants who achieve partial response (PR) or complete response (CR) only. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all lesions and normalization of tumor marker level. All lymph nodes (whether target or non-target) must be non-pathological in size (< 10mm short axis).
Time Frame: From first confirmed response to the date of the first documented tumor progression or death, up to approximately 48 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 96 | 46 | 26 | 18
Months | 11.01 [7.10 to NA] — Upper limit not calculated due to insufficient number of events | 37.68 [10.87 to NA] — Upper limit not calculated due to insufficient number of events | 16.51 [3.88 to 47.87] | 19.48 [6.28 to 20.57]

ADVERSE EVENTS:
Time Frame: SAEs and NSAEs: From first dose to 100 days post last dose (up to approximately 29 months). Participants were assessed for All-cause mortality from their first dose to study completion (up to approximately 56 months)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 55/106 | 29/52 | 15/28 | 20/25
Serious Adverse Events (participants affected / at risk) | 63/106 | 29/52 | 14/28 | 17/25
Other Adverse Events (participants affected / at risk) | 103/106 | 50/52 | 27/28 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=106) | Cohort 2 (N=52) | Cohort 3 (N=28) | Cohort 4 (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 1 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 5 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Cryptosporidiosis infection (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 2 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
CSF white blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 6 | 5 | 5
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=106) | Cohort 2 (N=52) | Cohort 3 (N=28) | Cohort 4 (N=25)
Anaemia (Blood and lymphatic system disorders) | 21 | 6 | 9 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 3 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 8 | 3 | 3 | 3
Hypothyroidism (Endocrine disorders) | 19 | 6 | 9 | 7
Dry eye (Eye disorders) | 2 | 3 | 0 | 0
Vision blurred (Eye disorders) | 7 | 2 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 17 | 7 | 6 | 7
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 24 | 14 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 45 | 19 | 11 | 9
Dry mouth (Gastrointestinal disorders) | 10 | 4 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 9 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 40 | 20 | 12 | 6
Stomatitis (Gastrointestinal disorders) | 9 | 5 | 1 | 3
Vomiting (Gastrointestinal disorders) | 24 | 12 | 3 | 1
Asthenia (General disorders) | 11 | 4 | 4 | 2
Chills (General disorders) | 10 | 6 | 3 | 0
Fatigue (General disorders) | 62 | 31 | 14 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 3 | 0 | 3
Oedema peripheral (General disorders) | 23 | 9 | 6 | 4
Pain (General disorders) | 4 | 3 | 0 | 1
Peripheral swelling (General disorders) | 4 | 0 | 2 | 0
Pyrexia (General disorders) | 13 | 9 | 3 | 2
Seasonal allergy (Immune system disorders) | 6 | 0 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 2 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 5 | 3 | 2 | 1
Pneumonia (Infections and infestations) | 6 | 2 | 1 | 2
Sinusitis (Infections and infestations) | 4 | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 4 | 2 | 2
Urinary tract infection (Infections and infestations) | 7 | 2 | 4 | 2
Fall (Injury, poisoning and procedural complications) | 10 | 2 | 1 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 2 | 0 | 3
Alanine aminotransferase increased (Investigations) | 15 | 5 | 2 | 1
Amylase increased (Investigations) | 15 | 6 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 14 | 6 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 10 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 21 | 3 | 5 | 7
Blood thyroid stimulating hormone decreased (Investigations) | 3 | 3 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 5 | 2 | 2 | 1
Lipase increased (Investigations) | 23 | 8 | 6 | 5
Weight decreased (Investigations) | 12 | 10 | 8 | 6
Weight increased (Investigations) | 7 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 26 | 14 | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 15 | 11 | 6 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 2 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 3 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 6 | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 1 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 1 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 4 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 1 | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 7 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 12 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 10 | 3 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 | 7 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 20 | 8 | 1 | 0
Headache (Nervous system disorders) | 19 | 12 | 5 | 2
Paraesthesia (Nervous system disorders) | 6 | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 1 | 1 | 0
Tremor (Nervous system disorders) | 2 | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 13 | 6 | 4 | 4
Confusional state (Psychiatric disorders) | 4 | 2 | 4 | 1
Depression (Psychiatric disorders) | 6 | 5 | 2 | 3
Insomnia (Psychiatric disorders) | 21 | 7 | 4 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 4 | 5
Haematuria (Renal and urinary disorders) | 3 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 11 | 7 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 8 | 3 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 11 | 9 | 5
Rash (Skin and subcutaneous tissue disorders) | 8 | 3 | 2 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 6 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 10 | 6 | 8
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 12 | 5 | 3 | 2
Hypertension (Vascular disorders) | 9 | 6 | 2 | 2
Hypotension (Vascular disorders) | 11 | 5 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02982954/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02982954/SAP_001.pdf